CLINICAL TRIAL: NCT03483454
Title: Improvement of Fitness and Health in Children With Obesity
Brief Title: Improvement of Fitness in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Pennsylvania American Academy of Pediatrics (Unknown)
Responsible Party: Principal Investigator, Marsha Novick, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00007398
Record Dates: First submitted 2018-02-08; First posted 2018-03-30 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Pediatric Obesity
Keywords: exercise, fitness, sleep, children, obesity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise classes (Experimental): This group of children and their parents will participate in an exercise class for 8 weeks.
  Interventions: Other: Exercise class
- Home exercise (Experimental): This group of children and their parents will participate in exercise at home for 8 weeks. This is currently the standard of care in the weight management clinic (advise to continue increasing activity at home). This group is considered the "control group."
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Exercise class — Same as above.
  Arms: Exercise classes
Other: Home exercise — Same as above.
  Arms: Home exercise

SUMMARY:
This study observes fitness level and health parameters in children ages 6-12 years old with obesity using an exercise class intervention.

DETAILED DESCRIPTION:
The purpose of this study is to improve physical fitness and health parameters in elementary-aged children who participate in an academic weight loss clinic. Patients and their parents are randomly assigned to either take exercise classes or to continue standard care (control group). Exercise classes are run at a local church 3 times a week for 8 weeks and children and parents are expected to participate. Parents are expected to follow similar dietary and exercise recommendations which are given to their children. Vitals, lab work and fitness testing are done on children at beginning, middle and end of the 6- month study. Vitals are done on parents at the beginning, middle and end of the study. Children are given Fitbits to record sleep patterns and daily physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Child must be a patient at the Penn State Hershey Children's Hospital Pediatric Multidisciplinary Weight Loss Program
* Child must be ages 6-12 years old

Exclusion Criteria:

* Lack of transportation to exercise classes
* Parents do not agree to participate in the exercise classes

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change in amount of Fitness in Obese Children as measured by daily physical activity via Fitbit | 8 weeks and 6 months
  measurement of amount of daily physical activity (in minutes) hours) as measured by daily physical activity via Fitbit
Program attendance by the child and parent in the exercise class arm | 8 weeks
  Class attendance will be taken at each class that is held 3x/week for 8 weeks
Change in intensity of daily activity in obese children | 8 weeks and 6 months
  measurement of intensity of daily activity measured by minutes of elevated heart rate via Fitbit
Change in sleep in obese children | 8 weeks and 6 months
  measurement of amount of sleep measured in hours via Fitbit

SECONDARY OUTCOMES:
Metabolic parameters of children with obesity: Body Mass Index (BMI) | 8 weeks and 6 months
  Height (in centimeters) and weight (in kilograms) will be measured by nurses at the Pediatric Weight Management Clinic. Height and weight will be combined to report Body Mass Index (BMI) in kg/m2
Metabolic parameters of children with obesity: blood pressure | 8 week and 6 months
  Blood pressure will be measured by nurses at the Pediatric Weight Management Clinic and reported as systolic blood pressure over diastolic blood pressure measured in millimeter of mercury (mmHg)
Metabolic parameters of children with obesity: resting heart rate | 8 weeks and 6 months
  Resting heart rate will be measured by nurses at the Pediatric Weight Management Clinic in beats per minute (BPM)
Metabolic parameters of children with obesity: Blood glucose (sugar) | 8 weeks and 6 months
  Lab work will be obtained to check fasting blood glucose in milligrams per deciliter (mg/dL)
Metabolic parameters of children with obesity: Cholesterol (Lipid Panel) | 8 weeks and 6 months
  Lab work will be obtained to check a fasting lipid panel, which includes total cholesterol (in milligrams per deciliter), LDL cholesterol (in milligrams per deciliter), HDL cholesterol (in milligrams per deciliter) and triglycerides (in milligrams per deciliter)
Metabolic parameters of children with obesity: Insulin level | 8 weeks and 6 months
  Lab work will be obtained to check fasting insulin level (in u International Units per milliliter)
Metabolic parameters of children with obesity: Hemoglobin A1c levels | 8 weeks and 6 months
  Lab work will be obtained to check hemoglobin A1c level (in percent of total hemoglobin)
Metabolic parameters of children with obesity: Liver Function Tests (LFTs) | 8 weeks and 6 months
  Lab work will be obtained to check liver function tests, including Aspartate Aminotransferase (in Units per liter) and Alanine Transaminase (in Units per liter)
Depression measurements in children with obesity | 8 weeks and 6 months
  The Center for Epidemiologic Studies Depression Scale (CES-DC) will be used to measure depressive symptoms in children. The scale ranges from 0-60; higher scores suggest greater prevalence of depressive symptoms
Motivation of children with obesity and their parents | 8 weeks and 6 months
  A survey will be distributed to the children and their parents at the beginning of their participation of the study, at the end of the 8-week exercise class period, and 6 months after enrollment. The survey will explore physical activity history and goals.
Fitness Testing of children with obesity | 8 weeks and 6 months
  All children in the study will be asked to complete a 6-minute fitness walking test (measured in feet) prior to the start of the study, at the end of the 8-week exercise class period, and 6 months after enrollment
Amount of sleep in children | daily for 6 months
  Amount of sleep will be measured in hours via Fitbit
Parental vital signs: blood pressure | 8 weeks and 6 months
  Blood pressure will be measured by nurses at the Pediatric Weight Management Clinic and reported as systolic blood pressure over diastolic blood pressure measured in millimeter of mercury (mmHg)
Parental vital signs: heart rate | 8 weeks and 6 months
  Resting heart rate will be measured nurses at the Pediatric Weight Management Clinic in beats per minute (BPM)
Parental vital signs: Body Mass Index (BMI) | 8 weeks and 6 months
  Height (in centimeters) and weight (in kilograms) will be measured by nurses at the Pediatric Weight Management Clinic. Height and weight will be combined to report Body Mass Index (BMI) in kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Marsha B Novick, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No